CLINICAL TRIAL: NCT05417035
Title: Pubertal Replacement In Boys Study Pubertal Induction in Boys With Delayed Puberty: Comparison Between Testosterone Enanthate and Testosterone Undecanoate Treatment.
Brief Title: Pubertal Replacement In Boys Study Nebido and Testoviron Depot Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NU-Hospital Organization, Sweden (Other)
Responsible Party: Principal Investigator, Martin Österbrand, Paediatrician, NU-Hospital Organization, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT nr 2012-002337-11
Record Dates: First submitted 2022-03-28; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Puberty Delayed
MeSH Terms: conditions — Puberty, Delayed | interventions — testosterone undecanoate

STUDY DESIGN:
Intervention Model Description: prospective open clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nebido (Experimental): i.m 250 mg/3months 2 injectionjs
  Interventions: Drug: Nebido
- Testoviron Depot (Active Comparator): i.m75mg/month 6 injections
  Interventions: Drug: Nebido

INTERVENTIONS:
Drug: Nebido — To evaluate if traditional treatment induces puberty similary to newer treatment
  Other Names: Testosteroneundecanoate

SUMMARY:
In this prospective open clinical study, Pubertal Replacement in Boys Study (PRIBS), boys 14-16 years with delayed puberty in terms of slow pubertal progression, were randomized to SoC treatment with TE: Testostoviron depot® 75 mg intramuscularly (i.m) / month (6 injections), or low dose TU: Nebido® 250mg i.m. / 3 months (2 injections). Our goal was to implement a study similar to clinical routine.

DETAILED DESCRIPTION:
Boys 14-16 years with pubertal delay were randomized to standard treatment with TE (Testosterone enanthat 75mg /month 6 injections)or newer treatment TU(Testosterone Undecanooat 250mg 2 injections 3 months apart) for pubertal induction. Our study PRIBS (pubertal replacement in boys study) was academically sponsored, monitored and approved by the medical products agency in Sweden. Between 2014 -08 and 2019-07 27 boys were randomized to treatment with TE (12 boys) or TU (15 boys). Testosterone levels were measured twice before study start and after 2,7,30,60,90,180 and 365 days. Boys with delayed puberty > 14 years with morning testosterone levels 0,5 - 3 Nmol/L and testicular volume ≤ 6 mL were included.Primary Outcome was testicular enlargement ≥ 8mL after 12 months. The new treatment was considered clinically similar if the treatment result were in the 80-125% interwall of the traditional group. Fishers exact chi square test was used for this analysis. Our intention was to recruit 20 boys in each armInformed consent was signed before study start by parents and assent by the boys. PRIBS was approved by the regional ethic committee 2012-09-14 Dnr 506-12 and approved by Union Drug Regulating Authorities Clinical Trials Database EudraCT nr 2012-002337-11 and the Swedish drug authorities (Läkemedelsverket) All study personal was trained in ICH GCP (good clinical practice).

ELIGIBILITY:
Inclusion Criteria:

* • Signed informed consent

  * Two morning testosterone values (07.30-09.00) of 1-3 nmol/L and at start < 4 mmol/L ¹
  * Testicular volume 4-6 mL bilaterally²

Exclusion Criteria:

* • Growth spurt

  * Untreated hypothyroidism, celiac disease or steroid medication
  * Training doses > 10 hours a week
  * Use of anabolic steroids or other drugs

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only for induction of puberty for boys (testosterone) For girls estradiol is used
Enrollment: 27 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Testicular Volume 8ml | 12 months after induction
  Evaluation by palpating the testicles

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and published
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Vill be shared after study published
Access Criteria: After the study has been published

REFERENCES:
- [Derived] Osterbrand M, Fors H, Norjavaara E. Pharmacological treatment for pubertal progression in boys with delayed or slow progression of puberty: A small-scale randomized study with testosterone enanthate and testosterone undecanoate treatment. Front Endocrinol (Lausanne). 2023 Apr 14;14:1158219. doi: 10.3389/fendo.2023.1158219. eCollection 2023. PMID 37124726

DOCUMENTS (1):
  • Statistical Analysis Plan (2013-01-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT05417035/SAP_000.pdf